CLINICAL TRIAL: NCT01750008
Title: The LUSTOR (Laparoscopic Uterine Sparing Techniques Outcomes and Reinterventions)Trial
Brief Title: Laparoscopic Uterine Sparing Techniques Outcomes and Reinterventions
Acronym: LUSTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acessa Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP-00-0018
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Uterine Fibroids; Myomas
Keywords: Symptomatic Uterine Fibroids; Menorrhagia; Heavy Bleeding; Myomas; Radiofrequency Ablation; RFA; Leiomyoma; Fibroids
MeSH Terms: conditions — Leiomyoma; Myoma; Menorrhagia | interventions — Uterine Myomectomy

STUDY DESIGN:
Intervention Model Description: Study compares two laparoscopic interventions for the treatment of symptomatic uterine fibroids.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Global Fibroid Ablation (Other): Global Fibroid Ablation
  Interventions: Procedure: Global Fibroid Ablation
- Laparoscopic Myomectomy (Other): Myomectomy via laparoscopy
  Interventions: Procedure: Myomectomy

INTERVENTIONS:
Procedure: Global Fibroid Ablation
  Other Names: Halt Procedure; Acessa Procedure
  Arms: Global Fibroid Ablation
Procedure: Myomectomy
  Arms: Laparoscopic Myomectomy

SUMMARY:
The purpose of this study is to compare the outcomes of two uterine-conserving treatment alternatives for symptomatic uterine fibroids: laparoscopic myomectomy (LM) and global fibroid ablation (GFA) using the Halt System. Laparoscopic ultrasound (LUS) is a standard step prior to the GFA procedure but has not been a standard step prior to LM. Incorporating laparoscopic ultrasound as a first step prior to both treatments allows the surgeon to have equal access to valuable imaging information and to plan treatment accordingly. By randomizing the subject immediately after laparoscopic ultrasound, selection bias toward one treatment or the other following the LUS is eliminated.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥ 18 years old and menstruating
* Have symptomatic uterine fibroids
* Have a uterine size ≤16 gestational weeks as determined by pelvic exam
* Have fibroids that are less than 10 cm in any diameter
* Desire uterine conservation
* Have had a normal Papanicolaou test (PAP smear) (i.e. PAP I or PAP II) at the latest pre-study examination and no longer than 36 months before study entry.
* Are willing and able to comply with all study tests, procedures, and assessment tools
* Are capable of providing informed consent.

Exclusion Criteria:

* Have contraindications for laparoscopic surgery and/or general anesthesia.
* Are expected to be high risk for, or are known to have, significant intra-abdominal adhesions (defined as adhesions that would require extensive dissection to mobilize and view all surfaces of the uterus)
* Patients requiring major elective concomitant procedures (e.g., hernia repair, hysteroscopic resection, endometrial ablation, uterine artery ligation, etc.) that could confound the results of the study
* Are pregnant or lactating
* Have taken any depot Gonadotropin-releasing hormone (GnRh agonist within three months prior to the screening procedures
* Have an implanted intrauterine or fallopian tube device for contraception that cannot or will not be removed at least ten days prior to treatment
* Have chronic pelvic pain not due to uterine fibroids
* Have known or suspected endometriosis or adenomyosis
* Have active or history of pelvic inflammatory disease
* Have a history of, or evidence of, gynecologic malignancy or pre-malignancy within the past five years
* Have had pelvic radiation
* Have a non-uterine pelvic mass over 3 cm
* Have a cervical myoma
* Have one or more completely intracavitary submucous fibroids (Type 0) or only Type 0/1 submucous fibroids that are better treated via hysteroscopic methods
* In the medical judgment of the investigator should not participate in the study
* Are not willing to be randomized to treatment.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Compare the mean time of hospitalization following laparoscopic treatment of fibroids by myomectomy or GFA | From admission to the duration of hospital stay, an expected average of 3 days
  Capture and compare hospitalization time expressed as the number of hours from induction of anesthesia to discharge from hospital.

SECONDARY OUTCOMES:
Compare and contrast post-treatment readmission and reintervention rate | Baseline and 3, 6, 12, 24, 36, 48, and 60 months post treatment
  Compare incidence of post discharge readmission within 1 month of procedure and rate of reintervention for fibroid-related symptoms up to 60 months post procedure
Compare and Contrast peri and post procedural safety including procedural blood loss and complications | Baseline and 3, 6, 12, 24, 36, 48, and 60 months post-treatment
  Compare intraoperative blood loss and rate of procedural-related complications up to 60 months post treatment
Compare and contrast recovery rate | Discharge from hospital up to an average of 5 weeks post treatment
  Compare how many days it takes to return-to-work and to normal activities of daily living.
Compare and Contrast post-treatment changes in fibroid symptom severity. | Baseline and 3, 6, 12, 24, 36, 48, and 60 months post-treatment
  Compare Baseline fibroid related symptoms to 3, 6, 12, 24, 36, 48 and 60 months post treatment
Compare and contrast post-treatment patient satisfaction | 3, 6, 12, 24, 36, 48, and 60 months post-treatment
  Compare the overall subject treatment outcome and satisfaction evaluation
Compare and Contrast post-treatment changes in menstrual status. | Baseline, 3, 6 ,12, 24, 36, 48, and 60 months post treatment
  Compare Baseline menstrual impact to 3, 6, 12, 24, 36, 48 and 60 months post treatment.
Compare and Contrast post-treatment changes concerning health-related quality-of-life. | Baseline, 3, 6 ,12, 24, 36, 48, and 60 months post treatment
  Compare Baseline general health outcome to 3, 6, 12, 24, 36, 48 and 60 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Brucker, MD, Principal Investigator — University of Tubingen
Locations (1):
- Tubingen University Hospital, Tübingen, Germany

REFERENCES:
- [Background] Spies JB, Coyne K, Guaou Guaou N, Boyle D, Skyrnarz-Murphy K, Gonzalves SM. The UFS-QOL, a new disease-specific symptom and health-related quality of life questionnaire for leiomyomata. Obstet Gynecol. 2002 Feb;99(2):290-300. doi: 10.1016/s0029-7844(01)01702-1. PMID 11814511
- [Background] Twijnstra AR, Kolkman W, Trimbos-Kemper GC, Jansen FW. Implementation of advanced laparoscopic surgery in gynecology: national overview of trends. J Minim Invasive Gynecol. 2010 Jul-Aug;17(4):487-92. doi: 10.1016/j.jmig.2010.03.010. Epub 2010 May 14. PMID 20471917
- [Background] Viswanathan M, Hartmann K, McKoy N, Stuart G, Rankins N, Thieda P, Lux LJ, Lohr KN. Management of uterine fibroids: an update of the evidence. Evid Rep Technol Assess (Full Rep). 2007 Jul;(154):1-122. PMID 18288885
- [Background] Holzer A, Jirecek ST, Illievich UM, Huber J, Wenzl RJ. Laparoscopic versus open myomectomy: a double-blind study to evaluate postoperative pain. Anesth Analg. 2006 May;102(5):1480-4. doi: 10.1213/01.ane.0000204321.85599.0d. PMID 16632830
- [Background] Parker WH, Iacampo K, Long T. Uterine rupture after laparoscopic removal of a pedunculated myoma. J Minim Invasive Gynecol. 2007 May-Jun;14(3):362-4. doi: 10.1016/j.jmig.2006.10.024. PMID 17478371
- [Background] Banas T, Klimek M, Fugiel A, Skotniczny K. Spontaneous uterine rupture at 35 weeks' gestation, 3 years after laparoscopic myomectomy, without signs of fetal distress. J Obstet Gynaecol Res. 2005 Dec;31(6):527-30. doi: 10.1111/j.1447-0756.2005.00331.x. PMID 16343253
- [Background] Mara M, Maskova J, Fucikova Z, Kuzel D, Belsan T, Sosna O. Midterm clinical and first reproductive results of a randomized controlled trial comparing uterine fibroid embolization and myomectomy. Cardiovasc Intervent Radiol. 2008 Jan-Feb;31(1):73-85. doi: 10.1007/s00270-007-9195-2. Epub 2007 Oct 18. PMID 17943348
- [Background] Manyonda IT, Bratby M, Horst JS, Banu N, Gorti M, Belli AM. Uterine artery embolization versus myomectomy: impact on quality of life--results of the FUME (Fibroids of the Uterus: Myomectomy versus Embolization) Trial. Cardiovasc Intervent Radiol. 2012 Jun;35(3):530-6. doi: 10.1007/s00270-011-0228-5. Epub 2011 Jul 20. PMID 21773858
- [Background] Munro MG, Critchley HO, Broder MS, Fraser IS; FIGO Working Group on Menstrual Disorders. FIGO classification system (PALM-COEIN) for causes of abnormal uterine bleeding in nongravid women of reproductive age. Int J Gynaecol Obstet. 2011 Apr;113(1):3-13. doi: 10.1016/j.ijgo.2010.11.011. Epub 2011 Feb 22. PMID 21345435
- [Background] Bushnell DM, Martin ML, Moore KA, Richter HE, Rubin A, Patrick DL. Menorrhagia Impact Questionnaire: assessing the influence of heavy menstrual bleeding on quality of life. Curr Med Res Opin. 2010 Dec;26(12):2745-55. doi: 10.1185/03007995.2010.532200. Epub 2010 Nov 3. PMID 21043553
- [Background] Hartung J, Knapp G. On tests of the overall treatment effect in meta-analysis with normally distributed responses. Stat Med. 2001 Jun 30;20(12):1771-82. doi: 10.1002/sim.791. PMID 11406840
- [Background] Levine DJ, Harris M, Berman JM, Macer J, Abbott K, Lee BB. Leiomyoma assessment by intra-abdominal ultrasound compared to preoperative ultrasound and preoperative magnetic imaging. J Minim Invasive Gynecol. 2011;18(suppl):S1.
- [Background] Moss JG, Cooper KG, Khaund A, Murray LS, Murray GD, Wu O, Craig LE, Lumsden MA. Randomised comparison of uterine artery embolisation (UAE) with surgical treatment in patients with symptomatic uterine fibroids (REST trial): 5-year results. BJOG. 2011 Jul;118(8):936-44. doi: 10.1111/j.1471-0528.2011.02952.x. Epub 2011 Apr 12. PMID 21481151
- [Background] U.S. Valuation of the EuroQoL EQ-5D Health States. December 2005. Agency for Healthcare Research and Quality, Rockville, MD. http://www.ahrq.gove/rice/EQ5Dproj.htm
- [Background] Chudnoff SG, Berman JM, Levine DJ, Harris M, Guido RS, Banks E. Outpatient procedure for the treatment and relief of symptomatic uterine myomas. Obstet Gynecol. 2013 May;121(5):1075-1082. doi: 10.1097/AOG.0b013e31828b7962. PMID 23635746
- [Background] Robles R, Aguirre VA, Argueta AI, Guerrero MR. Laparoscopic radiofrequency volumetric thermal ablation of uterine myomas with 12 months of follow-up. Int J Gynaecol Obstet. 2013 Jan;120(1):65-9. doi: 10.1016/j.ijgo.2012.07.023. Epub 2012 Oct 14. PMID 23073229
- [Background] Garza Leal JG, Hernandez Leon I, Castillo Saenz L, Lee BB. Laparoscopic ultrasound-guided radiofrequency volumetric thermal ablation of symptomatic uterine leiomyomas: feasibility study using the Halt 2000 Ablation System. J Minim Invasive Gynecol. 2011 May-Jun;18(3):364-71. doi: 10.1016/j.jmig.2011.02.006. PMID 21545960
- [Background] Guido RS, Macer JA, Abbott K, Falls JL, Tilley IB, Chudnoff SG. Radiofrequency volumetric thermal ablation of fibroids: a prospective, clinical analysis of two years' outcome from the Halt trial. Health Qual Life Outcomes. 2013 Aug 13;11:139. doi: 10.1186/1477-7525-11-139. PMID 23941588
- [Result] Brucker SY, Hahn M, Kraemer D, Taran FA, Isaacson KB, Kramer B. Laparoscopic radiofrequency volumetric thermal ablation of fibroids versus laparoscopic myomectomy. Int J Gynaecol Obstet. 2014 Jun;125(3):261-5. doi: 10.1016/j.ijgo.2013.11.012. Epub 2014 Feb 28. PMID 24698202
- [Result] Hahn M, Brucker S, Kraemer D, Wallwiener M, Taran FA, Wallwiener CW, Kramer B. Radiofrequency Volumetric Thermal Ablation of Fibroids and Laparoscopic Myomectomy: Long-Term Follow-up From a Randomized Trial. Geburtshilfe Frauenheilkd. 2015 May;75(5):442-449. doi: 10.1055/s-0035-1545931. PMID 26097247
- [Result] Kramer B, Hahn M, Taran FA, Kraemer D, Isaacson KB, Brucker SY. Interim analysis of a randomized controlled trial comparing laparoscopic radiofrequency volumetric thermal ablation of uterine fibroids with laparoscopic myomectomy. Int J Gynaecol Obstet. 2016 May;133(2):206-11. doi: 10.1016/j.ijgo.2015.10.008. Epub 2015 Dec 31. PMID 26892690
- [Result] Walter CB, Hartkopf AD, Schoeller D, Kraemer B, Neis F, Taran FA, Isaacson KB, Brucker SY, Hahn M. Ultrasound guided core needle biopsy prior to thermo ablative treatment of uterine tumors: first results. Arch Gynecol Obstet. 2018 Feb;297(2):387-392. doi: 10.1007/s00404-017-4590-7. Epub 2017 Nov 24. PMID 29177589
- [Derived] Berman JM, Guido RS, Garza Leal JG, Pemueller RR, Whaley FS, Chudnoff SG; Halt Study Group. Three-year outcome of the Halt trial: a prospective analysis of radiofrequency volumetric thermal ablation of myomas. J Minim Invasive Gynecol. 2014 Sep-Oct;21(5):767-74. doi: 10.1016/j.jmig.2014.02.015. Epub 2014 Mar 5. PMID 24613404